CLINICAL TRIAL: NCT00608569
Title: International Trial of Modified Directly Observed Therapy Versus Self-Administered Therapy for Participants With First Virologic Failure on a Non-Nucleoside Reverse Transcriptase Inhibitor-Containing Antiretroviral Regimen
Brief Title: Determining the Effects of Observed and Self-Administered Drug Regimens in HIV Infected Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ACTG A5234; 1U01AI068636 (NIH)
Record Dates: First submitted 2008-01-21; First posted 2008-02-06 (Estimated); Results first posted 2013-11-15 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-09

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; HIV Non-Nucleoside Reverse Transcriptase Inhibitors; HIV Protease Inhibitors; Viral Load; Virologic Failure
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir; lopinavir-ritonavir drug combination; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Tenofovir; Zidovudine; Emtricitabine

ARMS (2):
- mDOT arm (Experimental): Oral FTC/TDF+LPV/rtv or TDF+ZDV+LPV/rtv for 52 weeks. Modified directly observed therapy (mDOT) for the first 24 weeks and self-administration for the remaining 28 weeks.
  Interventions: Drug: Lopinavir/ritonavir; Drug: Emtricitabine/Tenofovir disoproxil fumarate; Drug: Tenofovir disoproxil fumarate; Drug: Zidovudine; Drug: Emtricitabine
- non-mDOT arm (Active Comparator): Oral FTC/TDF+LPV/rtv or TDF+ZDV+LPV/rtv for 52 weeks. Self-administration of the study treatment (non-mDOT) for 52 weeks.
  Interventions: Drug: Lopinavir/ritonavir; Drug: Emtricitabine/Tenofovir disoproxil fumarate; Drug: Tenofovir disoproxil fumarate; Drug: Zidovudine; Drug: Emtricitabine

INTERVENTIONS:
Drug: Lopinavir/ritonavir — Two tablets (200-mg lopinavir and 50 mg ritonavir in each tablet), taken orally twice daily
  Other Names: LPV/RTV; LPV/r; Kaletra
Drug: Emtricitabine/Tenofovir disoproxil fumarate — 200-mg emtricitabine and 300 mg tenofovir disoproxil fumarate in each tablet, taken orally once daily
  Other Names: FTC/TDF; Truvada
Drug: Tenofovir disoproxil fumarate — 300-mg tablet taken orally once daily
  Other Names: TDF; Viread
Drug: Zidovudine — 300-mg tablet taken orally twice daily
  Other Names: ZDV; Retrovir
Drug: Emtricitabine — 200-mg tablet taken orally once daily
  Other Names: FTC; Emtriva

SUMMARY:
Highly active antiretroviral therapy (HAART) has led to better health and survival rates among people with HIV/AIDS. The purpose of this study was to measure the effect of trained partner supervision when taking medication versus self-administered therapy in HIV infected participants. These participants have had their first virologic failure on a non-nucleoside reverse transcriptase inhibitor (NNRTI)-based HAART regimen and were starting a protease inhibitor (PI)-based HAART regimen at study entry.

DETAILED DESCRIPTION:
Poor adherence to HAART is usually associated with resistant virus. Poor adherence to HAART can have serious consequences, including limited treatment options for HIV infected individuals if they become infected with resistant HIV. The purpose of this study was to examine the effectiveness of modified directly observed therapy (mDOT) and compare it with the effectiveness of self-administered therapy (non-mDOT) in HIV infected individuals with first virologic failure on an NNRTI-based HAART regimen who were starting a PI-based HAART regimen at study entry.

mDOT was defined in this study as the daily observation of lopinavir/ritonavir (LPV/r) being taken on a regular basis. Observation consisted of an mDOT partner being present at the time the study participant took the observed dose. Half of the participants in this study were required to choose an mDOT partner to supervise adherence for the first 24 weeks of the study. Each mDOT partner completed the study-administered mDOT training program and was required to record all observed doses in an mDOT diary log. All participants and partners received health education through the study. Adherence was measured using Medication Event Monitoring System (MEMS) caps and self-report questionnaires.

This study lasted 52 weeks. Per protocol, participants were to be stratified according to their screening viral load and the proposed study treatment. The study treatment each participant received was based on their treatment history. At entry, participants were to start one of the two PI-based HAART regimens, either FTC/Tenofovir Disoproxil Fumarate (TDF) 200/300 mg once daily (QD) and Lopinavir/Ritonavir (LPV/RTV) 400/100 mg twice a day (BID) or TDF 300 mg QD and zidovudine (ZDV) 300 mg BID and LPV/RTV 400/100 mg BID. mDOT was used for the first 24 weeks of the study, followed by self-administration of study medications from week 25 to week 52. ZDV was not provided by the study. All enrolled participants except one who did not start study regimen initiated FTC/TDF and LPV/rtv after randomization. No participants started ZDV containing regimen on study. Thus, participants in this study were stratified by screening HIV-1 RNA only.

There were eight visits during the study. Medical and medication history, blood collection, and clinical assessment were required at all visits. A quality of life questionnaire and an adherence tools assessment were collected at most visits. For the mDOT arm, medication diary logs and mDOT partner monitoring were reviewed at most visits. An mDOT exit questionnaire and exit interview were required at the end of the study.

ELIGIBILITY:
Inclusion Criteria for Participants:

* HIV infected
* Have experienced or currently experiencing first baseline virologic failure on first NNRTI-based HAART regimen with no history of virologic failure on another regimen OR discontinued first NNRTI-based HAART regimen without the recommendations of clinicians and currently experiencing virologic failure with no history of virologic failure on another regimen. More information on this criterion can be found in the protocol.
* Confirmed virologic failure within 45 days of study entry
* Receiving one of the following NNRTI-based regimens for at least 16 weeks prior to study entry: ZDV+3TC+NVP, ZDV+3TC+EFV, d4T+3TC+NVP or d4T+3TC+EFV
* Able to identify a close friend, relative, or spouse who is willing to serve as a partner
* Intend to stay in current geographical area of residence for the duration of the study
* Agree to use LPV/rtv with MEMS caps and take the tablets out of the container only at dosing
* Willing to use acceptable forms of contraception
* Ability and willingness of participant or legal guardian/representative to give written informed consent.
* Required laboratory values obtained within 45 days prior to study entry.
* Negative serum or urine pregnancy test obtained within 48 hours prior to study entry for women of reproductive potential.

Inclusion Criteria for Partners:

* Not a participant
* Friend, family member, or spouse who knows of the participant's HIV status. Partners do not have to live with participants.
* Willing to attend a 1- to 2-hour taped training session prior to study entry
* Willing to attend study visits with participant at study screening; entry; and Weeks 4, 8, 12, 24, and 52
* Willing to directly observe participant taking at least one dose of LPV/rtv for at least 5 days per week for 24 weeks after stratification of participant
* Willing to act as a positive support for participant
* Willing to notify clinical staff of participant's nonadherence to study assigned regimen
* Willing to notify clinical staff if they are unable to provide mDOT for 2 weeks or more
* Willing to complete medication diary logs
* Willing to complete exit interview
* Agree to have their training session taped (if required).
* For mDOT arm, willing to discuss and decide with participants whether to continue mDOT after Week 24
* At least 18 years old
* Understand that participants have agreed to use LPV/RTV with MEMS caps and take the tablets out of the container only at dosing
* Ability and willingness to give written informed consent.
* No intention to relocate away from current geographical area of residence for the duration of study participation.

Exclusion Criteria for Participants:

* Use of any immunomodulator, HIV vaccine, or other investigational therapy within 45 days of study entry
* Prior treatment with any PI
* Previously diagnosed cancer other than basal cell carcinoma and cutaneous Kaposi's sarcoma
* Use of rifampin or rifabutin within 45 days of study entry or plan use of rifampin or rifabutin
* Requirement for taking any medications that are prohibited by this study. More information on this criterion can be found in the protocol.
* Known allergy to the study medications or their formulations
* Current drug or alcohol use that, in the opinion of the investigator, would interfere with the study
* Acute illness requiring hospitalization within 14 days of study entry
* Active tuberculosis (TB) infection
* Currently incarcerated
* Participation as a partner in this study
* Participation with no access to telephones
* Abnormal laboratory values
* Pregnant, breastfeeding, or intend to become pregnant

Exclusion Criteria for Partners:

* A participant in this study
* Participation as a partner to any other participant
* No access to telephones
* Currently incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 529 (Actual)
Dates: Start 2009-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gross, MD, MSCE, Study Chair — University of Pennsylvania; Alberto La Rosa, MD, Study Chair — Asociación Civil Impacta Salud y Educación, Peru
Locations (9):
- Gaborone Prevention/Treatment Trials CRS, Gaborone, Botswana
- Instituto de Pesquisa Clinica Evandro Chagas (12101), Rio de Janeiro, Brazil
- Les Centres GHESKIO CRS, Bicentenaire, Port-au-Prince, Haiti
- Peru (2):
  - San Miguel CRS, San Miguel, Lima region
  - Barranco CRS, Lima
- Wits HIV CRS, Johannesburg, Gauteng, South Africa
- JCRC CRS, Kampala, Uganda
- Kalingalinga Clinic CRS, Lusaka, Zambia
- UZ-Parirenyatwa CRS, Harare, Zimbabwe

REFERENCES:
- [Background] Bangsberg DR, Kroetz DL, Deeks SG. Adherence-resistance relationships to combination HIV antiretroviral therapy. Curr HIV/AIDS Rep. 2007 May;4(2):65-72. doi: 10.1007/s11904-007-0010-0. PMID 17547827
- [Background] Conway B. The role of adherence to antiretroviral therapy in the management of HIV infection. J Acquir Immune Defic Syndr. 2007 Jun 1;45 Suppl 1:S14-8. doi: 10.1097/QAI.0b013e3180600766. PMID 17525686
- [Background] Goggin K, Liston RJ, Mitty JA. Modified directly observed therapy for antiretroviral therapy: a primer from the field. Public Health Rep. 2007 Jul-Aug;122(4):472-81. doi: 10.1177/003335490712200408. PMID 17639650
- [Background] Pearson CR, Micek MA, Simoni JM, Hoff PD, Matediana E, Martin DP, Gloyd SS. Randomized control trial of peer-delivered, modified directly observed therapy for HAART in Mozambique. J Acquir Immune Defic Syndr. 2007 Oct 1;46(2):238-44. doi: 10.1097/QAI.0b013e318153f7ba. PMID 17693890
- [Derived] Mantshonyane L, Roy J, Levy MZ, Wallis CL, Bar K, Godfrey C, Collier A, LaRosa A, Zheng L, Sun X, Gross R. Participants Switching to Second-Line Antiretroviral Therapy with Susceptible Virus Display Inferior Adherence and Worse Outcomes: An Observational Analysis. AIDS Patient Care STDS. 2021 Dec;35(12):467-473. doi: 10.1089/apc.2021.0115. Epub 2021 Nov 16. PMID 34788110
- [Derived] De Boni RB, Zheng L, Rosenkranz SL, Sun X, Lavenberg J, Cardoso SW, Grinsztejn B, La Rosa A, Pierre S, Severe P, Cohn SE, Collier AC, Gross R. Binge drinking is associated with differences in weekday and weekend adherence in HIV-infected individuals. Drug Alcohol Depend. 2016 Feb 1;159:174-80. doi: 10.1016/j.drugalcdep.2015.12.013. Epub 2015 Dec 24. PMID 26774947
- [Derived] Gross R, Zheng L, La Rosa A, Sun X, Rosenkranz SL, Cardoso SW, Ssali F, Camp R, Godfrey C, Cohn SE, Robbins GK, Chisada A, Wallis CL, Reynolds NR, Lu D, Safren SA, Hosey L, Severe P, Collier AC; ACTG 5234 team. Partner-based adherence intervention for second-line antiretroviral therapy (ACTG A5234): a multinational randomised trial. Lancet HIV. 2015 Jan;2(1):e12-9. doi: 10.1016/S2352-3018(14)00007-1. Epub 2014 Dec 11. PMID 26424232

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited across 9 study sites (2 in Peru, one each in South Africa, Haiti, Uganda, Botswana, Zimbabwe, Brazil and Zambia) in the AIDS Clinical Trials Group system between April 2009 and September 2011.
Pre-assignment Details: Five hundred twenty nine subjects including participants and partners entered the study. Among the 529 subjects, 259 were participants, which included two participants with eligibility violations. Only the 257 eligible participants were included in the analyses. All participants started TDF/FTC +LPV/rtv and stratified by screening HIV-1 RNA only.
Period: Overall Study
Arm/Group | mDOT Arm | Non-mDOT Arm
Started | 129 | 128
Completed | 119 | 119
Not Completed | 10 | 9
Not completed — Death | 4 | 3
Not completed — Lost to Follow-up | 4 | 5
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Unable to adhere with study requirements | 0 | 1

BASELINE CHARACTERISTICS:
Population: Five hundred twenty nine subjects including participants and partners entered the study. Among the 529 subjects, 259 were participants, which include two participants with eligibility violations. Only the 257 eligible participants were included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | mDOT Arm | Non-mDOT Arm | Total
Number analyzed (Participants) | 129 | 128 | 257
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 127 | 123 | 250
  >=65 years | 1 | 5 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (9.7) | 39.4 (10.6) | 39.4 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 65 | 127
  Male | 67 | 63 | 130
Race/Ethnicity, Customized [Number; unit: participants]
  Black Non-Hispanic | 101 | 103 | 204
  Hispanic (regardless of race) | 27 | 25 | 52
  More than one race | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Haiti | 37 | 36 | 73
  Zambia | 4 | 5 | 9
  Botswana | 4 | 4 | 8
  Peru | 23 | 23 | 46
  Uganda | 25 | 25 | 50
  South Africa | 15 | 17 | 32
  Zimbabwe | 17 | 16 | 33
  Brazil | 4 | 2 | 6
CD4 Counts [Median (Inter-Quartile Range); unit: cells/mm3] — The baseline CD4 count is the average of screening and entry values.
  cells/mm3 | 164 [91 to 250] | 201 [97 to 292] | 179 [92 to 269]
CD4 Count Category [Number; unit: participants]
  0-50 cells/mm3 | 17 | 14 | 31
  51-100 cells/mm3 | 20 | 19 | 39
  101-200 cells/mm3 | 40 | 31 | 71
  201-350 cells/mm3 | 35 | 47 | 82
  351-500 cells/mm3 | 9 | 12 | 21
  >500 cells/mm3 | 8 | 5 | 13
Log10 HIV-1 RNA Viral Load [Median (Inter-Quartile Range); unit: log10 copies/mL] — The baseline HIV-1 RNA value is the result at study entry.
  log10 copies/mL | 4.2 [3.8 to 4.9] | 4.3 [3.8 to 4.9] | 4.3 [3.8 to 4.9]
HIV-1 RNA Viral Load Category [Number; unit: participants]
  <=400 copies/mL | 6 | 5 | 11
  401-999 copies/mL | 4 | 2 | 6
  1000-9999 copies/mL | 42 | 38 | 80
  10000-99999 copies/mL | 54 | 55 | 109
  100000-499999 copies/mL | 17 | 24 | 41
  >=500000 copies/mL | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Virologic Failure at or Prior to Week 48
Description: Confirmed virologic failure was defined as two successive HIV-1 RNA measurements at least 24 hours apart that were either:1) <1 log10 copies/mL below the baseline level and >400 copies/mL at the week 12 HIV-1 RNA evaluation (obtained at least 11 weeks after the date of the randomization) 2) >400 copies/mL at or after the week 24 HIV-1 RNA evaluation (obtained at least 23 weeks after the date of randomization). 3) subjects who discontinued the study follow-up for any reason other than study completion, including death, and who did so ≤50 weeks after randomization was considered to be a virologic failure. Number of participants experiencing or not experiencing virologic failure at or prior to week 48 was reported.
Time Frame: At or prior to Week 48
Population: Two hundred fifty seven eligible participants were included in the analysis. Intent to treat analysis was performed.
Measure: Number; unit: participants
Arm/Group | mDOT Arm | Non-mDOT Arm
Number analyzed (Participants) | 129 | 128
participants
  No Failure | 95 | 105
  Experienced Failure | 34 | 23
Statistical Analysis 1: Comparison: mDOT Arm vs Non-mDOT Arm; Fisher exact test (unstratified); Test type: Superiority or Other; p = 0.133, Fisher Exact — Results were considered to be statistically significant if p<0.05

2. Secondary Outcome: Confirmed Virologic Failure at or Prior to Week 24
Description: Confirmed virologic failure was defined as two successive HIV-1 RNA measurements at least 24 hours apart that were either:1) <1 log10 copies/mL below the baseline level and >400 copies/mL at the week 12 HIV-1 RNA evaluation (obtained at least 11 weeks after the date of the randomization) 2) >400 copies/mL at or after the week 24 HIV-1 RNA evaluation (obtained at least 23 weeks after the date of randomization). 3) subjects who discontinued the study follow-up for any reason other than study completion, including death, and who did so ≤30 weeks after randomization was considered to be a virologic failure. Number of participants experiencing or not experiencing virologic failure at or prior to week 24 was reported.
Time Frame: At or prior to Week 24
Population: Two hundred fifty seven eligible participants were included in the analysis. Intent to treat analysis was performed.
Measure: Number; unit: participants
Arm/Group | mDOT Arm | Non-mDOT Arm
Number analyzed (Participants) | 129 | 128
participants
  No Failure | 105 | 111
  Experienced Failure | 24 | 17

3. Secondary Outcome: CD4 Count at Follow-up Visits
Description: CD4 cell count (median, inter-quartile range)
Time Frame: At Weeks 4, 12, 24, 36, and 48
Measure: Median (Inter-Quartile Range); unit: cells/mm3
Arm/Group | mDOT Arm | Non-mDOT Arm
Number analyzed (Participants) | 129 | 128
cells/mm3
  Week 4 | 212 [129 to 309] | 219 [158 to 289]
  Week 12 | 225 [168 to 359] | 235 [174 to 337]
  Week 24 | 268 [177 to 382] | 266 [181 to 395]
  Week 36 | 281 [189 to 395] | 294 [214 to 418]
  Week 48 | 301 [198 to 432] | 347 [234 to 466]

4. Secondary Outcome: CD8 Count at Follow-up Visits
Description: CD8 cell count (median, inter-quartile range)
Time Frame: At week 4, 12, 24, 36, and 48
Measure: Median (Inter-Quartile Range); unit: cells/mm3
Arm/Group | mDOT Arm | Non-mDOT Arm
Number analyzed (Participants) | 129 | 128
cells/mm3
  Week 4 | 776 [557 to 1048] | 859 [557 to 1141]
  Week 12 | 895 [625 to 1155] | 916 [635 to 1290]
  Week 24 | 816 [586 to 1071] | 818 [547 to 1126]
  Week 36 | 787 [539 to 1034] | 833 [598 to 1131]
  Week 48 | 815 [566 to 1037] | 823 [573 to 1125]

5. Secondary Outcome: Time to First Grade 3 or 4 Lab Event
Description: 5th and 10th percentiles in weeks from randomization to first grade 3 or 4 lab event
Time Frame: 52 weeks since randomization
Population: Two hundred fifty seven eligible participants were included in the analysis. As-treated analysis was performed.
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | mDOT Arm | Non-mDOT Arm
Number analyzed (Participants) | 129 | 128
weeks
  5th percentile | 24 [1.3 to NA] — Not estimable as the upper limit for survival function at all weeks is above 95% | NA [12 to NA] — Not estimable as the estimates for survival function at all weeks is above 95%
  10th percentile | NA [12 to NA] — Not estimable as the estimates for survival function at all weeks is above 90% | NA [36.9 to NA] — Not estimable as the estimates for survival function at all weeks is above 90%

6. Secondary Outcome: Time to First Grade 3 or 4 Sign or Symptom
Description: 5th and 10th percentiles in weeks from randomization to first grade 3 or 4 sign or symptom
Time Frame: 52 weeks since randomization
Population: Two hundred fifty seven eligible participants were included in the analysis. As-treated analysis was performed.
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | mDOT Arm | Non-mDOT Arm
Number analyzed (Participants) | 129 | 128
weeks
  5th percentile | 13.7 [0 to 48] | 26.7 [0.3 to 48.9]
  10th percentile | NA [12 to NA] — Not estimable as the estimates for survival function at all weeks is above 90% | 48.9 [12 to NA] — Not estimable as the upper limit for survival function at all weeks is above 90%

7. Secondary Outcome: Time to First Grade 3 or 4 Lab or Sign/Symptom Event
Description: 5th and 10th percentiles in weeks from randomization to first grade 3 or 4 lab or sign/ symptom event
Time Frame: 52 weeks since randomization
Population: Two hundred fifty seven eligible participants were included in the analysis. As-treated analysis was performed.
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | mDOT Arm | Non-mDOT Arm
Number analyzed (Participants) | 129 | 128
weeks
  5th percentile | 6.4 [0 to 13.7] | 24 [0.3 to 32.1]
  10th percentile | 24 [4.4 to 48] | 32.6 [12 to NA] — Not estimable as the upper limit for survival function at all weeks is above 90%

8. Secondary Outcome: Adherence to Second Line HAART Regimen
Description: Number of participants with self-reported 100% adherence over the week prior to study visit
Time Frame: At weeks 4, 8, 12, 24, 36, 48 and 52
Population: Only the 257 eligible participants were included in the analysis. Self-reported adherence was collected face-to-face or by self-report on the Adherence/Quality of Life/Psychosocial Interview form. Only adherence to LPV/rtv was collected.
Measure: Number; unit: participants
Arm/Group | mDOT Arm | Non-mDOT Arm
Number analyzed (Participants) | 129 | 128
participants
  Week 4 | 105 | 117
  Week 8 | 108 | 115
  Week 12 | 114 | 116
  Week 24 | 107 | 116
  Week 48 | 103 | 109
  Week 52 | 104 | 109

ADVERSE EVENTS:
Time Frame: 52 weeks since randomization
Description: Expedited adverse event (AE) reporting followed Intensive Division of AIDS (DAIDS) Reporting Level, which included AEs resulting in death, congenital anomalies, fetal losses, significant disabilities, requiring hospitalization, and ≥grade 3 AEs (where grade 1=mild, 2=moderate, 3=severe, 4=life threatening/disabling, 5=death).
Arm/Group | mDOT Arm | Non-mDOT Arm
Serious Adverse Events (participants affected / at risk) | 6/129 | 7/128
Other Adverse Events (participants affected / at risk) | 94/129 | 98/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | mDOT Arm (N=129) | Non-mDOT Arm (N=128)
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 2 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 2 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | mDOT Arm (N=129) | Non-mDOT Arm (N=128)
Abdominal pain (Gastrointestinal disorders) | 4 | 9
Diarrhoea (Gastrointestinal disorders) | 16 | 18
Vomiting (Gastrointestinal disorders) | 6 | 9
Chest pain (General disorders) | 7 | 5
Pyrexia (General disorders) | 11 | 15
Urinary tract infection (Infections and infestations) | 4 | 10
Aspartate aminotransferase increased (Investigations) | 13 | 14
Blood alkaline phosphatase increased (Investigations) | 15 | 8
Blood bicarbonate abnormal (Investigations) | 9 | 8
Blood cholesterol (Investigations) | 0 | 7
Blood glucose increased (Investigations) | 14 | 9
Blood sodium decreased (Investigations) | 28 | 19
Blood sodium increased (Investigations) | 8 | 3
Haemoglobin decreased (Investigations) | 8 | 14
Neutrophil count decreased (Investigations) | 40 | 48
Weight decreased (Investigations) | 8 | 8
White blood cell count decreased (Investigations) | 24 | 21
Headache (Nervous system disorders) | 7 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights".